CLINICAL TRIAL: NCT00415246
Title: A Phase III, Single Arm, Multicentre Study to Evaluate the Efficacy and Safety of a Subcutaneous Four Months Sustained-release Formulation of Triptorelin, a Gonadotrophin Releasing Hormone Analogue in Patients With Prostate Cancer
Brief Title: Study to Evaluate a Subcutaneous Four Months Sustained-release Formulation of Triptorelin in Patients With Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The preliminary data do not support the expected sustainable blood levels of triptorelin for a duration of 4 months in all patients.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-55-52014-145; 2006-001511-30 (EudraCT Number)
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate; Therapeutics

INTERVENTIONS:
Drug: Triptorelin (Decapeptyl®) - Treatment 8 months (pivotal study) followed by a treatment extension of 8 months (extension study)

SUMMARY:
To identify the proportion of patients remaining medically castrated (testosterone level < 50 ng/dL) on Day 240 following two administrations of a 4-month sustained-release (SR) formulation of triptorelin.

ELIGIBILITY:
Inclusion Criteria:

* Patient must give written (personally signed and dated) informed consent before completing any study-related procedure, which means any assessment or evaluation that would not have formed part of the normal medical care of the patient
* Patient must be 18 years old or over
* Patient must have a histologically-confirmed diagnosis of locally advanced or metastatic prostate cancer or presenting a relapse after curative treatment which is amenable to androgen deprivation therapy
* Patient must have an estimated survival time of greater than 8 months according to the investigator's assessment

Exclusion Criteria:

* Patient at risk of a serious complication in the case of tumour flare (vertebral metastases threatening spinal cord compression or with significant obstructive uropathy)
* Patient who underwent a previous surgical castration
* Prostate cancer therapy within 2 months of baseline visit
* Patient with testosterone level below 150 ng/dL at screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-11; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with testosterone serum levels maintained below the castration threshold of 50 ng/dL. | Day 240

SECONDARY OUTCOMES:
Proportion of patients with testosterone serum levels maintained below the castration threshold of 50 ng/dL. | Day 120
Proportion of patients with testosterone serum levels maintained below the castration threshold of 20 ng/dL. | Day 120 and 240
Time to achieve castration in days post treatment (Tlag) | Day 35
Time to escape from castration (Texit) | Prior 4 months
Tlag and Texit confirmed by two consecutive measurements taken 1 week apart.
Duration of castration in days (Tcast) Changes in PSA levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (31):
- Belgium (5):
  - ULB Erasme, Brussels
  - Academisch Ziekenhuis Vrije Universiteit Brussel, Brussels
  - UCL St Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - UZ Gasthuisberg, Leuven
- France (12):
  - CHU Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Claude Huriez, Lille
  - Hôpital Edouard Herriot, Lyon
  - CHU Hôpital Salvator, Marseille
  - Hôtel Dieu, Nantes
  - Hôpital du Val de Grace, Paris
  - Centre Hospitalier Saint Louis, Paris
  - Hôpital Cochin, Paris
  - Hôpital Bichat, Paris
  - CHU Hôpital de la Miletrie, Poitiers
  - Hôpital Pontchaillou, Rennes
  - CHU Rangueil, Toulouse
- Latvia (3):
  - Olega Hublarova arsta prakse urologija, Daugavpils
  - Latvijas Onkologijas centre, Riga
  - Paula Stradina Kliniska Universitates slimnica, Riga
- Lithuania (3):
  - Kauno Medicinos Universitteto Klinikos, Kaunas
  - UAB 'Vilniaus onkourologijos-ginekologijos klinika, Vilnius
  - Vilniaus universiteto, Vilnius
- Poland (4):
  - Swietokrzyskie Centrum Onkologii, Kielce
  - NZOZ Specjalista Sp, z.o.o., Kutno
  - Centrum Onkologii Instytut im. M. Sklodowskiej-Curie, Warsaw
  - Akademicki Szpital Kliniczny, Wroclaw
- Hospital Gregorio Maranon, Madrid, Spain
- Ukraine (2):
  - Ivano Frankovsk State Medical University, Ivano-Frankivsk
  - Scientific Research Institute of Urology, Kiev
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom